CLINICAL TRIAL: NCT07183189
Title: A Randomized, Open-label, Multicenter, Phase III Study of SHR-A2009 Combined With Aumolertinib Versus Aumolertinib as First-line Treatment in Locally Advanced or Metastatic Non-Small Cell Lung Cancer With Epidermal Growth Factor Receptor (EGFR) Mutations
Brief Title: A Study of SHR-A2009 Combined With Aumolertinib Versus Aumolertinib for First-line Treatment in EGFR-mutated, Advanced or Metastatic NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2009-302
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- investigational treatment group：SHR-A2009 combined with Aumolertinib (Experimental)
  Interventions: Drug: SHR-A2009 ; Aumolertinib
- control group ：Aumolertinib (Active Comparator)
  Interventions: Drug: Aumolertinib

INTERVENTIONS:
Drug: SHR-A2009 ; Aumolertinib — SHR-A2009 administered intravenously, Aumolertinib administered orally.
  Arms: investigational treatment group：SHR-A2009 combined with Aumolertinib
Drug: Aumolertinib — Aumolertinib administered orally
  Arms: control group ：Aumolertinib

SUMMARY:
This study is a randomized, controlled, open-label, multicenter Phase III clinical trial designed to compare the efficacy and safety of SHR-A2009 combined with aumolertinib versus aumolertinib monotherapy in treatment-naïve subjects with EGFR-mutated, locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years (inclusive) at the time of signing informed consent, regardless of gender.
2. Subjects with histologically or cytologically confirmed locally advanced, metastatic, or recurrent non-small cell lung cancer, with EGFR mutations confirmed by tissue or blood specimens.
3. No prior systemic therapy for locally advanced, metastatic, or recurrent non-small cell lung cancer.
4. At least one measurable tumor lesion according to RECIST v1.1.
5. ECOG performance status of 0 or 1.
6. Expected survival time ≥12 weeks.
7. Adequate bone marrow and organ function.
8. Subjects must provide informed consent prior to the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Histologically or cytologically confirmed combined small cell lung cancer (SCLC), neuroendocrine carcinoma, sarcomatoid carcinoma, or carcinosarcoma components.
2. Subjects with a history of leptomeningeal metastasis, brainstem metastasis, or spinal cord metastasis.
3. Subjects with uncontrolled tumor-related pain, as determined by the investigator.
4. Clinically uncontrolled third-space fluid accumulation, as determined by the investigator.
5. Insufficient time interval between prior antitumor therapy and the first dose administration.
6. Major organ surgery or significant trauma within 4 weeks prior to the first dose of the study drug.
7. History of other malignancies within ≤5 years prior to the first dose.
8. Subjects with a history of interstitial lung disease, or imaging at screening suggestive of suspected interstitial lung disease; or other moderate to severe pulmonary diseases severely affecting lung function.
9. Severe cardiovascular or cerebrovascular diseases.
10. Any severe or uncontrolled ocular lesions that, in the physician's judgment, may increase the patient's safety risk.
11. Refractory nausea, vomiting, chronic gastrointestinal diseases, etc.
12. Severe infections within 4 weeks prior to the first dose.
13. Subjects with arterial/venous thromboembolic events within 6 months prior to the first dose of the study drug.
14. Active tuberculosis infection.
15. History of immunodeficiency, including positive HIV test.
16. Active hepatitis B or hepatitis C.
17. Prior allogeneic hematopoietic stem cell transplantation or organ transplantation.
18. History of severe allergic reactions to aumolertinib or other monoclonal antibodies, or hypersensitivity to any component of SHR-A2009.
19. Known history of alcohol or drug dependence or drug abuse.
20. Psychiatric disorders or poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2032-11 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by BICR according to RECIST v1.1 | Up to approximately 38 months

SECONDARY OUTCOMES:
overall survival (OS) | Up to approximately 60 months
Progression Free Survival(PFS by investigator) | Up to approximately 38months
Duration of response(DoR，by BICR and investigator ) | Up to approximately 38 months
Disease control rate（DCR，by BICR and investigator） | Up to approximately 38 months
Incidence of AEs | from Day1 to 40 days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided